CLINICAL TRIAL: NCT06839729
Title: Addressing Parental Tobacco Use in Somali Immigrant Families: Adapting an Evidence-based Intervention in Pediatric Primary Care
Brief Title: Addressing Parental Tobacco Use in Somali Immigrant Families: Adapting an Evidence-Based Intervention in Primary Care
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMCH-2024-33169
Record Dates: First submitted 2025-01-23; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEASE+ (Experimental): Clinician- and/or staff-delivered messaging and tobacco cessation resources to Somali parents who smoke
  Interventions: Behavioral: CEASE+

INTERVENTIONS:
Behavioral: CEASE+ — The intervention will be delivered by the clinician to smoking parents who attend the office visit and to smoking parents not present at the visit via resources sent home with a non-smoking parent. If the smoking parent is present in clinic, the intervention consists of a brief, clinician- delivered motivational intervention that includes messaging around the risks of household smoking, verbal recommendation for establishing home/car smoke-free rules, a printed prescription for nicotine replacement therapy and quitline information, and messaging on the benefits of cessation and a quitline referral. If the smoking parent is not present in clinic, the intervention will include clinician-delivered messaging to the non-smoking parent to share CEASE+ resources with the parent who smokes and an invitation for the parent who smokes to participate in a single call delivered by a culturally-/linguistically-congruent community health worker to connect them to CEASE+ resources.

SUMMARY:
This study will modify an existing evidence-based parental tobacco cessation intervention (the Clinical Effort Against Secondhand Smoke Exposure, or CEASE) delivered in pediatric primary care clinics to address shared tobacco use determinants and barriers to smoking cessation treatment among Somali Americans, an immigrant population facing significant combustible tobacco use disparities.

DETAILED DESCRIPTION:
Smoking is a significant and growing concern within U.S. Somali immigrant populations, who experience unique barriers to accessing and using tobacco treatments developed for the general population. Household smoking exposes Somali families to second- and thirdhand smoke with related negative health consequences and influences children's tobacco use beliefs and future behaviors. This study will modify and then pilot test an existing evidence-based parental tobacco cessation intervention (the Clinical Effort Against Secondhand Smoke Exposure, or CEASE) delivered in pediatric primary care clinics to address shared tobacco use determinants and barriers to smoking cessation treatment among Somali Americans. This new intervention, CEASE+, will increase access to and utilization of tobacco cessation treatment for Somali parents through brief clinician- and staff-delivered messaging and tobacco cessation resources. The project will take place in two phases. In phase 1, the investigators will modify the existing intervention to develop CEASE+ by conducting focus groups with Somali parents who smoke and non-smokers who live with adults who smoke and with the help of a community advisory board. In phase 2, we will conduct a pilot study of the new intervention, CEASE+, with Somali parents in 2 pediatric primary care clinics (n=50 parents who smoke). Primary outcomes will include feasibility and acceptability of CEASE+ intervention components and study procedures.

Secondary outcomes will include cigarette smoking abstinence and total tobacco abstinence at 3 months and changes in cigarette smoking heaviness between baseline and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* self-reported 1 st or 2 nd generation Somali identity
* parent or legal guardian at least one pediatric patient within the MHF system
* self-reported use of combustible cigarettes (even a puff) in the past 30 days
* access to a telephone

Exclusion Criteria:

Clinician or staff participant:

* Inability or unwillingness to participate in implementing CEASE+
* Employees or students of the research team

Parent participant:

* Having participated in Aim 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of parents who received motivational intervention | baseline
  The proportion of parents who report receipt of this tobacco cessation resource (dichotomous - yes/no)
Proportion of parents who received a verbal recommendation for smoke- free home/care rules | baseline
  The proportion of parents who report receipt of this tobacco
  cessation resource (dichotomous - yes/no)
Proportion of parents who received nicotine replacement therapy (NRT) | baseline
  The proportion of parents who report receipt of this tobacco
  cessation resource (dichotomous - yes/no)
Proportion of parents who received a quitline referral | baseline
  The proportion of parents who report receipt of this tobacco
  cessation resource (dichotomous - yes/no)
Percent completion of adapted protocol content | baseline
  The mean percent completion of adapted protocol participants
Mean duration of telephone call | baseline
  The mean duration of the coaching call (minutes)
Change in parental smoker utilization of NRT | baseline, 3months
  The change in the proportion of parental smoker utilization of NRT between baseline and 3 month follow up
Change in parental smoker utilization of quitline referrals | baseline, 3 months
  The change in the proportion of parental smoker utilization of quitline referrals between baseline and 3 month follow
Survey completion rate verification | baseline, 3 months
  The proportion of questions completed relative
Mean duration of telephone survey | baseline, 3 months
  The mean duration of telephone survey calls at baseline and 3 month follow up
Participation rate of recruitment (approached) | baseline
  The proportion of participants recruited over the proportion of
  participants approached
Participation rate of recruitment (eligible) | Baseline
  The proportion of participants recruited over the proportion of participants who are eligible based on a positive household
Retention of participants for follow-up | 3 month follow up
  The proportion of participants who remain in the study at the 3 month follow up time point
Abstinence verification participation | 3 month followup
  The proportion of participants reporting abstinence at 3 months who submit a sample for iCO biochemical verification
Mean participant satisfaction with CEASE+ materials | baseline
  Mean participant satisfaction score measured with 5-point Likert scale score (0 = strongly dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, 4=strongly satisfied)
Mean participant satisfaction with in-clinic motivational intervention | baseline
  Mean participant satisfaction score measured with 5-point Likert scale score (0 = strongly dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, 4=strongly satisfied)
Mean participant satisfaction with telephone- call delivered motivational intervention | baseline
  Mean participant satisfaction score measured with 5-point Likert scale score (0 = strongly dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, 4=strongly satisfied)
Mean participant satisfaction with CEASE+ messaging | baseline
  Mean participant satisfaction score measured with 5-point Likert scale score (0 = strongly dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, 4=strongly satisfied)
Mean participant satisfaction with study procedures (baseline) | Baseline
  Mean participant satisfaction score measured with 5-point Likert scale score (0 = strongly dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, 4=strongly satisfied)
Mean participant satisfaction with study procedures (follow up) | 3 month followup
  Mean participant satisfaction score measured with 5-point Likert scale score (0 = strongly dissatisfied, 1=dissatisfied, 2=neutral, 3=satisfied, 4=strongly satisfied)

SECONDARY OUTCOMES:
Parental cigarette smoking abstinence | 3 month follow up
  7-day point prevalence abstinence of combustible
Total tobacco product abstinence | 3 month follow up
  7-day point prevalence abstinence of all tobacco products including shisha, cigars, chew, e-cigarettes
Change in cigarette smoking heaviness | baseline and 3 month follow up
  Change in the heaviness of cigarette smoking score from baseline to 3 month follow up using the Heaviness of Smoking index measure
Change in the frequency of other tobacco use | baseline and 3 month follow up
  Change from baseline and 3 months in the proportion of parental smoker reported use of other forms of tobacco as a combined measure (i.e., e-cigarettes, hookah, cigars, etc.)
Change in the presence of smoke-free home/car rules | baseline and 3 month follow up
  Change from baseline to 3 month follow up in the proportion of participants who report the presence of smoke-free home/car rules using a 2-item measure "House Rules about

CONTACTS AND LOCATIONS:
Overall Officials: April Wilhelm, MD, MPH, Principal Investigator — University of Minnesota